CLINICAL TRIAL: NCT02903017
Title: Local Administration of Tranexamic Acid in Upper Gastrointestinal Hemorrhage: A Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: Local Administration of Tranexamic Acid in Upper Gastrointestinal Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nurettin Özgür Doğan, M.D., Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIA 2016/196
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Gastrointestinal Hemorrhage; Tranexamic Acid; Emergency Department; Antifibrinolytic Agents
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid 5% (Active Comparator): Tranexamic acid 5%, 2000 mg (40 mL) in 60 mL normal saline (0.9%) solution (total 100 mL)
  Interventions: Drug: Tranexamic acid 5%
- Placebo (Placebo Comparator): 0.9% normal saline solution (total 100 mL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid 5% — Via nasogastric tube, 100 mL
  Arms: Tranexamic acid 5%
Drug: Placebo — Via nasogastric tube, 100 mL
  Arms: Placebo

SUMMARY:
Upper gastrointestinal hemorrhage is a frequently diagnosis in emergency departments. Although new drugs and endoscopic techniques were easily applied in various settings in this condition, the role of local administered therapies such as antifibrinolytic agents remain unclear. The investigators aimed to compare standard therapy (proton pump inhibitors, endoscopic treatments etc.) and standard therapy + local administered tranexamic acid in upper gastrointestinal hemorrhage in a double-blind, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with upper gastrointestinal hemorrhage to the ED
* Patients older than 18 years
* Patients who agree to participate the study by reading and signing the informed consent form

Exclusion Criteria:

* Patients younger than 18 years
* Patients who do not agree to participate the study
* Documented or declared allergy to tranexamic acid
* Upper gastrointestinal hemorrhage secondary to trauma
* Upper gastrointestinal hemorrhage secondary to esophageal varices
* Patients who cannot undergo to endoscopy for any reason
* History for thromboembolic disease
* Patients with renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Mortality | One month
  In- or out of hospital mortality
Re-bleeding | One month
  Recurrent upper gastrointestinal hemorrhage
Endoscopic intervention need | One month
Surgical intervention need | One month
ED revisit | One month

SECONDARY OUTCOMES:
Length of stay in the hospital | One month
Administered blood products in the ED | One month
Adverse reactions | One month
  Thromboembolic events, anaphylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin Özgür Doğan, M.D., Assoc. Prof., Principal Investigator — Kocaeli University, Faculty of Medicine
Locations (1):
- Kocaeli University, Faculty of Medicine, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Hawkey GM, Cole AT, McIntyre AS, Long RG, Hawkey CJ. Drug treatments in upper gastrointestinal bleeding: value of endoscopic findings as surrogate end points. Gut. 2001 Sep;49(3):372-9. doi: 10.1136/gut.49.3.372. PMID 11511559
- [Background] Bergqvist D, Dahlgren S, Hessman Y. Local inhibition of the fibrinolytic system in patients with massive upper gastrointestinal hemorrhage. Ups J Med Sci. 1980;85(2):173-8. doi: 10.3109/03009738009179185. PMID 7018048
- [Background] Cormack F, Chakrabarti RR, Jouhar AJ, Fearnley GR. Tranexamic acid in upper gastrointestinal haemorrhage. Lancet. 1973 Jun 2;1(7814):1207-8. doi: 10.1016/s0140-6736(73)90525-4. No abstract available. PMID 4122561